CLINICAL TRIAL: NCT04040738
Title: Comparative Measurement of the Concentration of Blood Somatostatin and Fatty Amid Acids in Upper Extremity Trauma Surgery Under General and Regional Anesthesia
Brief Title: Plasma Concentration of Somatostatin and Endocannabinoids After GA and RA in Upper Extremity Trauma Surgery
Acronym: SECsGRUES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7726
Record Dates: First submitted 2019-06-05; First posted 2019-08-01 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pain; Arm Injury
MeSH Terms: conditions — Pain, Postoperative; Arm Injuries

STUDY DESIGN:
Intervention Model Description: Study participants n=25 in the S-GA, n=25 in the S-RA, n=25 in the H-GA, and n=25 in the H-RA Groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The labour analyst, the investigator, the statistician is unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper extremity surgery under general anaesthesia (Active Comparator): Fentanyl 2 mcg/kg iv, propofol 2 mg/kg iv induction, 1MAC sevoflurane maintenance
  Interventions: Procedure: Upper extremity surgery under general anaesthesia
- Upper extremity surgery under regional anaesthesia (Active Comparator): Bupivacaine brachial plexus block 0.4 ml/kg of 0.33% solution
  Interventions: Procedure: Upper extremity surgery under regional anaesthesia

INTERVENTIONS:
Procedure: Upper extremity surgery under general anaesthesia — Forearm, wrist and hand surgery after fentanyl and propofol induction of anaesthesia, with sevoflurane maintenance
  Arms: Upper extremity surgery under general anaesthesia
Procedure: Upper extremity surgery under regional anaesthesia — Forearm, wrist and hand surgery under brachial plexus block with 0.4 ml/kg of 0.33% bupivacaine solution Other Names: Marcaine 5 mg/ml Astra Zeneca OGYI-T 6496/14
  Arms: Upper extremity surgery under regional anaesthesia

SUMMARY:
The application of RA can decrease the central sensitization and chronic pain after trauma surgery. The plasma concentrations of somatostatin and fatty acid amides were not studied up to this time in this kind of settings, so investigators believe that this is the first work that shows how upper extremity nerve blockade changes the plasma concentration of somatostatin and fatty acid amides in upper limb surgery in trauma patients.

DETAILED DESCRIPTION:
Total of 100 American Society of Anesthesiologist (ASA) I-III, adult patients scheduled to elective or emergency trauma surgery of hand/forearm or shoulder are planned to be randomly allocated to general anaesthesia (GA) or ultrasound-guided (UG) brachial plexus block (BPB) group, in this randomized-prospective study after approval by the University Research Ethics Board, Pécs University Medical School, Hungary. All of the patients will receive detailed information about the planned BPB or GA techniques and surgeries, then written informed consents will be obtained. Study participants are planned to be assigned randomly into 4 groups (Shoulder GA; Shoulder RA; Hand/forearm GA; Hand/forearm RA).

Standardized UG Axillary-supraclavicular (AX-SC) approach to the BP is planned to be performed under sterile conditions, or standardized GA with propofol IV, fentanyl IV, and 1 MAC (minimal alveolar concentration) sevoflurane, by experienced anesthesiologists.

Blood samples will be taken at 0-time point (straight before the administration of BP injection or the induction of GA) and straight after the surgery. The collected serum samples are stored at -70 °C for a maximum of two weeks prior to analysis. Qualitative and quantitative determination of endocannabinoids and corticosteroids is performed by supercritical fluid chromatography coupled with tandem mass spectrometry after salting-out assisted liquid-liquid microextraction. For somatostatin measurement, the samples are immediately supplemented with aprotinin (20µl/ml blood sample; Gordox 10 KIU/ml (Kallikrein Inhibitor Unit/ml), Richter Gedeon Budapest, Hungary) and transported for centrifugation on ice. The pellet is discarded, and the plasma is stored at -80⁰C until further processing. The somatostatin concentration of the plasma sample is determined with both ELISA (CEA592Hu, Cloud-Clone Corp., Wuhan, PRC) and radioimmunoassay. The results are collected and analyzed.

Demographic data, vital parameters, and verbal numeric rate of pain intensity are collected prior to and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* upper extremity fracture
* surgery of hand/forearm or upper arm
* unpremedicated patients
* scheduled for elective or emergency trauma

Exclusion Criteria:

* psycho-mental conditions interfering with consent or assessment
* the patient refused to participate
* preexisting chronic pain condition
* daily analgesic or sedative or steroid consumption
* sedative or analgesic premedication
* pre-existing neuro-endocrine disorders
* antecedent cancer
* advanced liver or kidney disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Somatostatin concentration in plasma | 0-6 hours after surgery
  Plasma concentrations of somatostatin straight after and 6 hours after surgery.

SECONDARY OUTCOMES:
Endocannabinoid concentrations in plasma | 0-6 hours
  Plasma concentrations of endocannabinoids straight after and 6 hours after surgery.
Corticosteroid concentrations in plasma | 0-6 hours
  Plasma concentrations of corticosteroids straight after and 6 hours after surgery.

OTHER OUTCOMES:
Postoperative pain intensity: verbal numeric rate scale | 0-24 hours
  Postoperative pain intensity in a 0-10 point verbal numeric rate scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Almasi, PhD.Habil., Study Chair — University of Pecs, Medical School, Clinical Centre, Pain Medicine Dept.of Anesth Int Care; Zsofia Kriszta, MD., Principal Investigator — University of Pecs, Medical School, Clinical Centre, Dept.of Anesth Int Care
Locations (1):
- University of Pécs, Medical School, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No